CLINICAL TRIAL: NCT02490410
Title: A Double-blind Randomized Controlled Study About the Effects of Whey Protein Intervention on Body Composition and Muscular Function in the Elderly With Sacropenia
Brief Title: Effects of Whey Protein Intervention on Body Composition and Muscle Function in the Elderly With Sacropenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huilian Zhu (Other)
Responsible Party: Sponsor-Investigator, Huilian Zhu, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CNS-YILI2014-034
Record Dates: First submitted 2015-06-30; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- whey protein (Experimental): 2 x 10g whey protein per day orally for 6 months
  Interventions: Dietary Supplement: protein supplement
- whey protein+soy protein (Other): 10g whey protein + 10g soy protein per day orally for 6 months
  Interventions: Dietary Supplement: protein supplement
- soy protein (Other): 2 x 10g soy protein per day orally for 6 months
  Interventions: Dietary Supplement: protein supplement

INTERVENTIONS:
Dietary Supplement: protein supplement

SUMMARY:
The purpose of this study is to compare the effects of different dose of whey protein intervention(in a daily dose of 0g, 10g, 20g) on lean body mass,body fat composition and muscular function state in the elderly with sacropenia.

ELIGIBILITY:
Inclusion Criteria:

* People aged over 65 years.
* Usual gait speed less than 0.8m/s.
* Willing to participate in the study, consume the test product and perform all measurements.

Exclusion Criteria:

* nervous system disease.
* Other diseases with movement disorder such as stroke,fracture,arthritis.
* people who unconsciousness and can not complete questionnaire
* long-term regular use of protein and antioxidant.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
lean body mass | up to 6 months
  At baseline, 3 and 6 months, investigators will use DXA to examine lean body mass and body fat composition
muscular function state | up to 6 months
  At baseline, 3 and 6 months, investigators will use the Short Physical Performance Battery (SPPB) to test muscular function state

SECONDARY OUTCOMES:
plasma amino acid spectrum, especially branched chain amino acid spectrum | up to 6 months
  At baseline and 6 months, blood samples will be drawn and plasma amino acid spectrum, especially branched chain amino acid spectrum will be tested